CLINICAL TRIAL: NCT02249715
Title: Pilot Study for Development of a Monitoring Set-up and Algorithm Using Functional MRI (fMRI) and EEG for Prediction of Response to Repetitive Deep Transcranial Magnetic Stimulation (rDTMS) for Patients With Parkinson's Disease
Brief Title: Development of a Monitoring Set-up and Algorithm Using Functional MRI (fMRI) and EEG for Prediction of Response to Repetitive Deep Transcranial Magnetic Stimulation (rDTMS) for Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Brainsway (Industry); ElMindA Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-1293-14-OC-CTIL
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson
Keywords: Parkinson; TMS; BNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rDTMS (Experimental)
  Interventions: Device: Brainsway Multiway deep TMS device (two channels)

INTERVENTIONS:
Device: Brainsway Multiway deep TMS device (two channels)

SUMMARY:
* To characterize physiological biomarkers of positive response to rDTMS using EEG and functional MRI (fMRI) in patients with PD.
* To develop a set-up and algorithm for neurophysiological monitoring for PD patients using EEG and fMRI in patients treated by rDTMS.
* To integrate rDTMS stimulation with monitoring techniques with the ultimate goal of providing closed-loop feedback where monitoring informs the stimulation

DETAILED DESCRIPTION:
PD Patients aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria will be treated by an established rDTMS protocol will be monitored before, during and after rDTMS using quantitative EEG and brain network analysis and fMRI while performing a series of cognitive and motor tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD patients aged 40-75 years;
2. Hoehn and Yahr stages II to IV
3. Patients on stable antiparkinsonian therapy for 1 month
4. Right hand dominance with right afflicted side.

Exclusion Criteria:

1. Participation in current clinical study or clinical study within 30 days prior to this study.
2. Subject has an atypical parkinsonian syndrome or secondary parkinsonism (e.g., due to drugs, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease or other degenerative disease)
3. Patients with significant psychiatric symptoms or history.
4. Patients with psychotic symptoms or active depressive symptoms
5. Treatment with neuroleptics.
6. Beck depression inventory (BDI) score <14
7. Mini Mental status examination (MMSE) score <25
8. History of migraine or frequent or severe headaches.
9. Significant sensory deficits, e.g., deafness or blindness History of head injury or neurosurgical interventions.
10. Subjects who have concomitant epilepsy, a history of seizure/s, heat convulsions or history of epilepsy in first degree relative.
11. History of any metal in the head (outside the mouth).
12. The presence of cochlear implants
13. Known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
14. Subjects with an unstable medical disorder.
15. Current drug abuse (including Cannabis) or alcoholism.
16. Pregnancy or not using a reliable method of birth control.
17. Patients with severe tremor or dyskinesia

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 3 month